CLINICAL TRIAL: NCT02189070
Title: What Patients Really Want - Patient Preferences Regarding Annual Follow-up After Medical Interventions: The PAPAYA Study
Brief Title: The PAtient Preference Analysis of Yearly Follow-up After PCI (PAPAYA)
Acronym: PAPAYA
Status: Completed | Type: Observational
Sponsor: Thorax Centrum Twente (Other)
Responsible Party: Principal Investigator, Clemens von Birgelen, Professor, Thorax Centrum Twente
Other Study IDs: K13-28
Record Dates: First submitted 2014-07-11; First posted 2014-07-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
Keywords: Follow-up; Percutaneous coronary intervention; Patient preference; DUTCH PEERS; TWENTE
MeSH Terms: conditions — Coronary Artery Disease; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Responders: Responding participants
- Non-responders: Non-responding participants

SUMMARY:
The purpose of this study is to determine the preference of patients regarding the approach for follow-up after percutaneous coronary intervention (PCI) procedures. We hypothesize that patients prefer questionnaires for annual follow-up assessment when compared to telephone or email.

DETAILED DESCRIPTION:
Rationale: Assessment and reporting of long-term clinical follow-up after medical interventions is essential for transparency of medical care and its quality improvement. However follow-up adherence is a serious challenge in clinical trials. Taking the patient preference of the mode of follow-up into account is likely to enhance trial adherence, reduce withdrawals, and facilitate a longer follow-up duration. No data on patient preference of annual follow-up have been reported.

Objective: To investigate the patient preference of approach to obtain follow-up information after percutaneous coronary intervention (PCI)

Study design: Single-center, prospective, observational registry

Study population: All patients enrolled in the percutaneous coronary intervention studies TWENTE trial (a broad study population reflecting real-world PCI patients) and DUTCH PEERS trial (an all-comers population), who were treated at Thoraxcentrum Twente in Enschede between June 2008 and May 2012

Intervention: All subjects will receive a questionnaire with questions regarding their preference with regards to the approach of acquiring follow-up information after PCI.

Main study endpoints:

* The primary endpoint is the patient preference on how to be approached for annual follow-up after PCI procedures.
* Secondary endpoints include

  1. least preferred approach of follow-up
  2. the preferred number of follow-up moments per year
  3. the from the patients' perspective maximum acceptable number of questions to be answered
  4. the assessment of potential relationships between the most and least preferred approach of assessment and patient age, gender urgency of PCI treatment, and history of previous revascularizations

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the TWENTE trial and DUTCH PEERS trial (an all-comers population, who were treated at Thoraxcentrum Twente in Enschede between June 2008 and May 2012

Exclusion Criteria:

* Patients who had withdrawn their consent for participation in the TWENTE and DUTCH PEERS trials, respectively. Patients who passed away during follow-up could obviously not be approached for further questioning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in the percutaneous coronary intervention (PCI) studies TWENTE trial (a broad study population reflecting real-world PCI patients) and DUTCH PEERS trial (an all-comers populatoin), who were treated at Thoraxcentrum Twente in Enschede between June 2008 and May 2012
Sampling Method: Non-Probability Sample
Enrollment: 2566 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Assessment of preferred approach for annual follow-up after PCI | 1 year

SECONDARY OUTCOMES:
Least preferred approach for follow up | 1 year
Maximum acceptable number of questions to be answered | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clemens von Birgelen, MD,PhD,Prof, Principal Investigator — Thorax Centrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Netherlands

REFERENCES:
- [Derived] Kok MM, von Birgelen C, Lam MK, Lowik MM, van Houwelingen KG, Stoel MG, Louwerenburg JH, de Man FH, Hartmann M, Doggen CJ, van Til JA, IJzerman MJ. Patient preference regarding assessment of clinical follow-up after percutaneous coronary intervention: the PAPAYA study. EuroIntervention. 2016 Apr 20;11(13):1487-94. doi: 10.4244/EIJY15M10_06. PMID 26465376